CLINICAL TRIAL: NCT03060018
Title: Agreement of Transcutaneous Partial Oxygen and Carbon Dioxide Pressure With Arterial and Capillary Blood Gas Values. A Single Centre Prospective Non-randomized Trial in Critically Ill Neonates.
Brief Title: Transcutaneous Partial Oxygen and Carbon Dioxide Pressures Compared With Blood Gas Values
Acronym: OxiVenT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vera Bernet, MD (Other)
Responsible Party: Sponsor-Investigator, Vera Bernet, MD, Senior Consultant Pediatric Intensive Care, University Children's Hospital, Zurich
Organization: University Children's Hospital, Zurich (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KISPI-OXIVENT 3.0
Record Dates: First submitted 2017-02-11; First posted 2017-02-23 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All included patients (Experimental): All included patients will undergo the intervention of transcutaneous sensor placement
  Interventions: Device: Sentec (SenTec) Digital Monitoring System with OxiVenT Sensor

INTERVENTIONS:
Device: Sentec (SenTec) Digital Monitoring System with OxiVenT Sensor — The sensor will be attached to four anatomical positions (thoracic left and right; abdominal left and right), starting with the left thoracic position followed by 4-hourly clockwise position rotation. In case of severe oedema, the ear lobes will be used as anatomical measurement sites and changes to the contralateral ear lobe are made every 4 hours.

SUMMARY:
Partial blood oxygen and carbon dioxide pressures obtained in critical ill neonates by transcutaneous sensors will be compared to respective values obtained by medically indicated arterial and capillary blood gas analyses. The influence of blood withdrawal method, sensor operational temperature and application time, presence of cyanotic heart malformations and/or intra or extra cardiac right to left shunt, vasoactive drugs, elevated non-conjugated bilirubin, and skin and soft tissue oedema, skin colour and perfusion conditions will be elucidated as well as sensor's safety. Study duration will be 48 hours with sensors applied and additional 4 hours of further surveillance for thermal injury.

ELIGIBILITY:
Inclusion Criteria:

* Late premature or term birth newborn infants (34 0/7 until 43 6/7 weeks gestational age (GA)).
* Age between first day of life and 43 6/7 weeks postmenstrual age.
* Ability of care taker to understand verbal and written instructions and informed consent in German.

Exclusion Criteria:

* Care taker unable or unwilling to give written informed consent in German.
* Care taker not understanding German and without a family member able to translate.
* Written informed consent cannot be obtained for any other reason.

Max Age: 10 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 113 (Actual)
Dates: Start 2017-08-17 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Bias and precision of the transcutaneous oxygen and carbon dioxide measurements | 52 hours
  Agreement of transcutaneous measurements with capillary and arterial blood gas values at two operational sensor temperatures (42 and 43°C).

SECONDARY OUTCOMES:
Agreement of partial transcutaneous oxygen and carbon dioxide pressures with arterial and capillary values in children with echocardiographically determined congenital cyanotic heart disease and/or intra or extra cardiac right to left shunt | 52 hours
Bias and precision of oxygen and carbon dioxide transcutaneous measurements under the influence of vasoactive drugs (Adrenalin, Noradrenalin, Dopamine, Dobutamine, Vasopressin, Milrinone) | 52 hours
Bias and precision of oxygen and carbon dioxide transcutaneous measurements under the influence of elevated indirect bilirubin | 52 hours
Bias and precision of the oxygen and carbon dioxide transcutaneous measurements over time at one anatomical site with determination of technical drift and physiological drift | 52 hours
Bias and precision of transcutaneous partial oxygen and carbon dioxide pressure measurements in patients with skin and soft tissue oedema | 52 hours
Bias and precision of transcutaneous partial oxygen and carbon dioxide pressure measurements with changing peripheral perfusion | 52 hours
Bias and precision of transcutaneous partial oxygen and carbon dioxide pressure measurements with different skin colour types | 52 hours
Safety of OxiVenT sensor: Appearance of signs of thermal injury (redness, blisters, necrosis) under application of transcutaneous sensor temperatures of 42 and 43°C | 52 hours
  While operated at sensor temperatures of 42 and 43°C, the skin will be closely observed for any kind of thermic tissue damage

CONTACTS AND LOCATIONS:
Overall Officials: Vera Bernet, Prof, MD, Principal Investigator — University of Zurich
Locations (1):
- University Children's Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baumann P, Gotta V, Adzikah S, Bernet V. Accuracy of a Novel Transcutaneous PCO2 and PO2 Sensor with Optical PO2 Measurement in Neonatal Intensive Care: A Single-Centre Prospective Clinical Trial. Neonatology. 2022;119(2):230-237. doi: 10.1159/000521809. Epub 2022 Feb 4. PMID 35124680